CLINICAL TRIAL: NCT05068947
Title: Safety, Tolerability, and Pharmacokinetic Study of Single Ascending Dose of GV101 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Graviton Bioscience Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBS-101
Record Dates: First submitted 2021-09-26; First posted 2021-10-06 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2021-09

CONDITIONS: Phase 1
Keywords: Healthy; Adult; Volunteers

STUDY DESIGN:
Intervention Model Description: 3:1 GV101 (study drug) to placebo. (1:1 for sentinel 2 subjects and 5:1 thereafter)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study drug: GV101 (Experimental): 400 mg (10 mL liquid), 800 mg (20 mL liquid), 1600 mg (40mL liquid) of GVS101 will be administered once, orally to subjects in the treatment group, cohort 5 to 7.
  Interventions: Drug: GV101
- Placebo (Placebo Comparator): Matched placebo control 400 mg (10 mL liquid), 800 mg (20 mL liquid), 1600 mg (40mL liquid) of GVS101 will be administered once, orally to subjects in the control group, cohort 5 to 7.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GV101 — GV101 administered once orally.
  Arms: Study drug: GV101
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
This is a single center Phase 1, placebo-controlled, randomized, double blind, first-in-human (FIH), sequential single ascending dose (SAD) study.

DETAILED DESCRIPTION:
GBS-101 is a single center Phase 1, placebo-controlled, randomized, double blind, first-in-human (FIH), sequential single ascending dose (SAD) study to evaluate the safety, tolerability and PK of GV101 in healthy subjects. 8 healthy subjects wills be enrolled cohorts 5 - 7 cohorts of the study. Cohorts 1-4 were previously completed with a tablet form of the study drug at 50 mg, 100 mg, 200 mg, and 400 mg. Planned cohorts 5 - 7 will be dosed 400 mg (liquid), 800 mg (liquid), 1600 mg (liquid) or matched placebo.. Participants will be randomized in a 3:1 ratio, 1:1 for 2 sentinel subjects and 5: 1 GV101 drug to matching placebo thereafter. Subjects in each cohort will receive a single oral dose of GV101 or matching placebo under fasting conditions. A staggered schedule will be used for each dose level, where 2 sentinel subjects (1 active and 1 placebo) will be dosed first, with the remaining 6 subjects (5 active and 1 placebo) dosed at least 24 hours after the sentinel subjects.

This study of GV101 will provide safety, tolerability, and plasma pharmacokinetic data in healthy individuals. The PK component will characterize the PK of GV101 to inform dosing and may help to correlate exposures treatment-related AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to

   a) communicate in English or Spanish b) provide written informed consent to take part in the study c) be available for all visits and able and willing to comply with all study procedural requirements
2. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥ 18 and ≤ 55 years of age, with BMI > 18.5 and < 30.0 kg/m2 and body weight within 50 kg and 100 kg for males and 45 kg and 100 kg for females.
3. Healthy, as defined by:

   a) The absence of clinically significant illness or surgery within 4 weeks of dosing. Subjects vomiting within 24 hours before the first study drug administration will be carefully evaluated for possible illness/disease and inclusion is at the discretion of the Investigator.

   b) The absence of clinically significant history and condition of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease
4. Women (sex at birth) Pre-menopausal women (not post-menopausal: absence of menses for at least 12 months and a medical history consistent with menopause) engaging in heterosexual sex that could lead to pregnancy must be willing to use an effective method of contraception for 4 weeks prior to taking the study drug, throughout the study and until 30 days following the last study drug intake: Acceptable methods are:

   • condom used together with another barrier method (diaphragm or cervical cap with spermicide), hormonal method started at least 8 weeks before dosing, or an IUD in place for at least 8 weeks

   • sterilization of participant or partner (male vasectomized for at least 6 months)
5. Men (sex at birth) Heterosexually active men are required to use an effective method of contraception for 4 weeks prior to taking the study drug, throughout the study and until 90 days following the last study drug intake: Acceptable methods are:

   • condom used together with another barrier method (diaphragm or cervical cap with spermicide), hormonal method started at least 8 weeks before dosing, or an IUD in place for at least 8 weeks

   • sterilization of participant or partner (male vasectomized for at least 6 months)
6. Male subjects must commit to not donate sperm until at least 90 days following study drug administration even if vasectomized.
7. Male subjects of a pregnant partner must use a condom from study drug administration until 90 days afterwards, even if the male partner has been vasectomized.

   -

Exclusion Criteria:

1. Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for hepatitis B, hepatitis C, or HIV found during medical screening
2. Evidence of hepatic or renal impairment including ALT and AST above 1.5 x ULN, total bilirubin above 1.5 x ULN, or creatinine above 1.5 x ULN.
3. Positive urine cotinine or positive urine drug screen at screening or baseline
4. History of anaphylaxis, or history of moderate or worse allergic reaction to oral drug excipients
5. History of clinically significant gastrointestinal diseases or surgery which might influence drug absorption
6. Positive pregnancy test at screening or baseline
7. Received a COVID-19 vaccine within 7 days of the baseline visit
8. Positive COVID-19 PCR test at screening or baseline
9. Clinically significant ECG abnormalities (QTcF ≥ 450 ms)
10. Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening or baseline. In cases of abnormal vital signs, tests can be repeated at the investigator's discretion.
11. History of substance abuse within 6 months before admission (with the exception of medically indicated marijuana), including alcohol
12. Use of an investigational drug or device or participation in an investigational study within 30 days prior to admission
13. Use of medications in the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

    1. Prescription medications taken within 14 days prior to dosing
    2. Over-the-counter and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals amino acids, essential fatty acids, and protein supplements used in sports) taken within 7 days prior to dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily)
    3. Depot injection or implant of any drug within 3 months prior to dosing
    4. Use of any drugs known to induce or inhibit hepatic drug metabolism (including St. John's Wort [hypericin]) within 30 days prior to dosing.
14. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to dosing
15. Breast feeding
16. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Treatment emergent AEs | Up to day 7.
  Number of TEAEs grade 2 or higher per Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.

SECONDARY OUTCOMES:
GV101 plasma levels will be quantified for PK analysis | Cohort 5 -7: pre-dose and 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72 hrs post dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: No